CLINICAL TRIAL: NCT01009905
Title: Registry of Patients Being Treated With Norditropin®, Recombinant Human Growth Hormone
Brief Title: An Observational Study (Registry) Assessing Treatment Outcomes and Safety for Children and Adults Who Are Prescribed Norditropin® (Human Growth Hormone)
Acronym: ANSWER
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: HGH-2149; U1111-1111-1168 (Other: WHO); NCT00615953 (obsolete NCT alias)
Record Dates: First submitted 2009-11-05; First posted 2009-11-09 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Growth Hormone Disorder; Pituitary Dwarfism; Hypopituitarism
MeSH Terms: conditions — Dwarfism, Pituitary; Hypopituitarism | interventions — Human Growth Hormone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — Safety and effectiveness data collection in connection with the use of Norditropin® (somatropin) in daily clinical practice

SUMMARY:
This study is conducted in the United States of America (USA). The aim of this observational study is to collect data concerning the treatment outcomes and safety for children and adults who are prescribed Norditropin®. Specific objectives include: 1) developing models defining the relationship of Norditropin dose to changes in insulin-like growth factor (IGF-I) and treatment outcomes, accounting for independent factors such as age, gender and puberty and 2) determining the relative predictive values of peak growth hormone (GH) and IGF-I levels and other factors before treatment to clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained
* Children or adult patients treated with Norditropin® for an appropriate condition as prescribed by their physician

Exclusion Criteria:

* Patients not being treated with Norditropin®
* Patients who have discontinued treatment with Norditropin®
* Known or suspected allergy to Norditropin® or related products
* Contraindications for somatropin treatment consistent with the Prescribing Information for Norditropin®

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients from both general and specialty practice settings, existing and new users of growth hormones, who have been deemed appropriate to receive Norditropin® as part of routine out-patient care by the prescribing physician.
Sampling Method: Non-Probability Sample
Enrollment: 22960 (Actual)
Dates: Start 2002-06-24 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
Change in height, measured as the height standard deviation score (HSDS), from the measurement made by the physician at study entry to the most recent clinic observation, end of GH treatment, de-registration, or change of clinic. | measurement made by physician at study entry, annually, or more frequently at physician discretion during the study.
Change in waist/hip circumference ratio for adult patients | measurement made by physician at study entry, annually, or more frequently at physician discretion during the study

SECONDARY OUTCOMES:
Short-term: Height, Height velocity, Height velocity standard deviation score (SDS), predicted adult height, height SDS for bone age, Proportion achieving height SDS > -2 at end of observational duration period | measurement made by physician at study entry, annually, or more frequently at physician discretion during the study.
Final Height (or Adult height), Final Height SDS, near-adult height, near-adult height SDS, Final Height - Target Height, Final height - predicted adult height, height age | measurement made by physician at study entry, annually, or more frequently at physician discretion during the study.
Final Height SDS - Target Height SDS, Final height SDS - predicted adult height SDS | measurement made by physician at study entry, annually, or more frequently at physician discretion during the study.
Proportion achieving HSDS of more than -2 at final height | measurement made by physician at study entry, annually, or more frequently at physician discretion during the study.
Weight, waist circumference, and hip circumference for adult patients | measurement made by physician at study entry, annually, or more frequently at physician discretion during the study

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), MD, Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Plainsboro, New Jersey, United States

REFERENCES:
- [Result] Ross JL, Lee PA, Gut R, Germak J. Attaining genetic height potential: Analysis of height outcomes from the ANSWER Program in children treated with growth hormone over 5 years. Growth Horm IGF Res. 2015 Dec;25(6):286-93. doi: 10.1016/j.ghir.2015.08.006. Epub 2015 Aug 22. PMID 26363846
- [Result] Lee PA, Savendahl L, Oliver I, Tauber M, Blankenstein O, Ross J, Snajderova M, Rakov V, Pedersen BT, Christesen HT. Comparison of response to 2-years' growth hormone treatment in children with isolated growth hormone deficiency, born small for gestational age, idiopathic short stature, or multiple pituitary hormone deficiency: combined results from two large observational studies. Int J Pediatr Endocrinol. 2012 Jul 12;2012(1):22. doi: 10.1186/1687-9856-2012-22. PMID 22788856
- [Result] Hoybye C, Savendahl L, Christesen HT, Lee P, Pedersen BT, Schlumpf M, Germak J, Ross J. The NordiNet(R) International Outcome Study and NovoNet(R) ANSWER Program(R): rationale, design, and methodology of two international pharmacoepidemiological registry-based studies monitoring long-term clinical and safety outcomes of growth hormone therapy (Norditropin(R)). Clin Epidemiol. 2013 Apr 26;5:119-27. doi: 10.2147/CLEP.S42602. Print 2013. PMID 23658497
- [Result] Savendahl L, Blankenstein O, Oliver I, Christesen HT, Lee P, Pedersen BT, Rakov V, Ross J. Gender influences short-term growth hormone treatment response in children. Horm Res Paediatr. 2012;77(3):188-94. doi: 10.1159/000337570. Epub 2012 Apr 12. PMID 22508317
- [Derived] Rohrer TR, Kotnik P, Miller BS, Kelepouris N, Olsen AH, Pietropoli A, Polak M, Blair J. Better growth outcomes in GH-deficient children treated younger than 2 years of age. Endocr Connect. 2025 Sep 23;14(9):e250493. doi: 10.1530/EC-25-0493. Print 2025 Sep 1. PMID 40919719
- [Derived] Backeljauw P, Blair JC, Ferran JM, Kelepouris N, Miller BS, Pietropoli A, Polak M, Savendahl L, Verlinde F, Rohrer TR. Early GH Treatment Is Effective and Well Tolerated in Children With Turner Syndrome: NordiNet(R) IOS and Answer Program. J Clin Endocrinol Metab. 2023 Sep 18;108(10):2653-2665. doi: 10.1210/clinem/dgad159. PMID 36947589
- [Derived] Biller BMK, Hoybye C, Carroll P, Gordon MB, Birkegard AC, Kelepouris N, Nedjatian N, Weber MM. Pregnancy outcomes in women receiving growth hormone replacement therapy enrolled in the NordiNet(R) International Outcome Study (IOS) and the American Norditropin(R) Studies: Web-Enabled Research (ANSWER) Program. Pituitary. 2021 Aug;24(4):611-621. doi: 10.1007/s11102-021-01138-3. Epub 2021 Mar 12. PMID 33709288
- [Derived] Savendahl L, Polak M, Backeljauw P, Blair JC, Miller BS, Rohrer TR, Hokken-Koelega A, Pietropoli A, Kelepouris N, Ross J. Long-Term Safety of Growth Hormone Treatment in Childhood: Two Large Observational Studies: NordiNet IOS and ANSWER. J Clin Endocrinol Metab. 2021 May 13;106(6):1728-1741. doi: 10.1210/clinem/dgab080. PMID 33571362
- [Derived] Angulo M, Abuzzahab MJ, Pietropoli A, Ostrow V, Kelepouris N, Tauber M. Outcomes in children treated with growth hormone for Prader-Willi syndrome: data from the ANSWER Program(R) and NordiNet(R) International Outcome Study. Int J Pediatr Endocrinol. 2020 Nov 10;2020(1):20. doi: 10.1186/s13633-020-00090-6. PMID 33292530
- [Derived] Miller BS, Ross J, Ostrow V. Height outcomes in children with growth hormone deficiency and idiopathic short stature treated concomitantly with growth hormone and aromatase inhibitor therapy: data from the ANSWER program. Int J Pediatr Endocrinol. 2020;2020:19. doi: 10.1186/s13633-020-00089-z. Epub 2020 Oct 6. PMID 33042202
- [Derived] Weber MM, Gordon MB, Hoybye C, Jorgensen JOL, Puras G, Popovic-Brkic V, Molitch ME, Ostrow V, Holot N, Pietropoli A, Biller BMK. Growth hormone replacement in adults: Real-world data from two large studies in US and Europe. Growth Horm IGF Res. 2020 Feb;50:71-82. doi: 10.1016/j.ghir.2019.09.002. Epub 2019 Oct 26. PMID 31972476
- [Derived] Savendahl L, Polak M, Backeljauw P, Blair J, Miller BS, Rohrer TR, Pietropoli A, Ostrow V, Ross J. Treatment of Children With GH in the United States and Europe: Long-Term Follow-Up From NordiNet(R) IOS and ANSWER Program. J Clin Endocrinol Metab. 2019 Oct 1;104(10):4730-4742. doi: 10.1210/jc.2019-00775. PMID 31305924
- [Derived] Rose SR, Reeves G, Gut R, Germak J. Attention-Deficit/Hyperactivity Disorder Medication Treatment Impact on Response to Growth Hormone Therapy: Results from the ANSWER Program, a Non-Interventional Study. J Pediatr. 2015 Dec;167(6):1389-96. doi: 10.1016/j.jpeds.2015.08.036. Epub 2015 Sep 26. PMID 26394822
- [Derived] Lee PA, Ross J, Germak JA, Gut R. Effect of 4 years of growth hormone therapy in children with Noonan syndrome in the American Norditropin Studies: Web-Enabled Research (ANSWER) Program(R) registry. Int J Pediatr Endocrinol. 2012 Jun 8;2012(1):15. doi: 10.1186/1687-9856-2012-15. PMID 22682146
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com